CLINICAL TRIAL: NCT03416985
Title: A Comparative Study of Electric Toothbrushes for the Efficacy Plaque Removal and the Effect on Plaque Accumulation and Gingivitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joan PiAnfruns, DMD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-001622
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Dental Plaque Induced Gingivitis; Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Manual Toothbrush (Active Comparator): Patients will be asked to use a manual toothbrush for 30 days
  Interventions: Device: Oral B Healthy Clean Manual Toothbrush
- Sonic Toothbrush (Active Comparator): Patients will be asked to use a sonic toothbrush for 30 days
  Interventions: Device: BURST Sonic Oral Care
- Pulsating Toothbrush (Active Comparator): Patients will be asked to use a pulsating toothbrush for 30 days
  Interventions: Device: Philipps Sonicare DiamondClean 300 Series

INTERVENTIONS:
Device: Oral B Healthy Clean Manual Toothbrush — Manual Toothbrush
  Arms: Manual Toothbrush
Device: BURST Sonic Oral Care — Electric sonic toothbrush
  Arms: Sonic Toothbrush
Device: Philipps Sonicare DiamondClean 300 Series — Electric pulsating toothbrush
  Arms: Pulsating Toothbrush

SUMMARY:
It is well accepted that the greatest contributor to the health of the periodontium and dentition is regular and thorough dental plaque removal, typically by means of adequate toothbrushing. Although patients are typically informed about the risks of substandard oral hygiene and the contributing factors in oral/dental disease by dental professionals, research has shown that an undesirably high proportion of adults find thorough toothbrushing with a standard manual toothbrush to achieve a plaque-free state challenging, as evidenced by high worldwide levels of gingivitis and/or periodontitis.

DETAILED DESCRIPTION:
The purpose of this study is to clinically evaluate the plaque removal efficacy of two electric powered toothbrushes after a single use, as well as the effect on plaque accumulation and gingivitis after 14 days and 30 days period. Simultaneously, a comparison against a manual toothbrush will be made.

Study design: randomised, single blinded, parallel.

After the screening procedure and based on inclusion requirements, all subjects will receive oral prophylaxis (T0) to ensure a baseline of 0 Plaque Index (PI) prior to the first appointment (T1). The subjects will be instructed not to use a tooth brush or any mechanical cleaning device until the initial PI and Gingival Indexes (GI) are taken at 24 hours after T0.

The subjects will be randomized into 3 groups, and the will be provided one of the three evaluated toothbrushes, as well as toothpaste. All subjects will be using identical toothpaste and will receive oral hygiene instructions based on the manufacturer's recommendations.

At T1 initial GI and PI will be taken prior to brushing followed by a second PI reading immediately after the first use of the power driven toothbrush.

The subjects will be instructed to brush twice a day for a period of 2 minutes (following the programmed toothbrush timer) and refrain from using dental floss, tooth pick or any mechanical oral hygiene aid for the period of the study.

On the second visit at 14 days (T2) and third visit at 30 days (T3), additional GI and PI readings will be taken and data will be recorded. All measurements and clinical examinations will be performed by a single blinded examiner. Evaluation on teeth will be made on six teeth #3,7,12,19,23 and 28 (mesio-buccal, buccal, disto-buccal and mesio-lingual, lingual, disto-lingual) following the Silness-Loe Index.

ELIGIBILITY:
Inclusion Criteria:

1. Good overall health
2. At least 20 teeth present, not including 3rd Molars
3. Non-smoker

Exclusion Criteria:

1. Poor manual dexterity or mentally handicap;
2. Presence of removable intra-oral prosthesis
3. Current orthodontic therapy
4. Severe Periodontal condition or caries teeth in need of immediate attention
5. Pregnant women
6. Subjects that use medications that may effect oral health
7. No Systemic diseases/conditions such as diabetes mellitus, heart disease.
8. Use of plaque inhibiting toothpaste, mouthwash, interdental flossing in the period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA School of Dentistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulsating Toothbrush: Patients were asked to use a pulsating toothbrush for 30 days Philipps Sonicare DiamondClean 300 Series: Electric pulsating toothbrush
- Sonic Toothbrush: Patients were asked to use a sonic toothbrush for 30 days
  BURST Sonic Oral Care: Electric sonic toothbrush
- Manual Toothbrush: Patients were asked to use a manual toothbrush for 30 days Oral B Healthy Clean Manual Toothbrush: Manual Toothbrush
Period: Overall Study
Arm/Group | Pulsating Toothbrush | Sonic Toothbrush | Manual Toothbrush
Started | 30 | 30 | 30
Completed | 28 | 30 | 24
Not Completed | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsating Toothbrush | Sonic Toothbrush | Manual Toothbrush | Total
Number analyzed (Participants) | 28 | 30 | 24 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 24 | 82
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 14 | 49
  Male | 12 | 11 | 10 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 24 | 82

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: plaque index as evaluated by Silness-Loe Index: index recording both soft debris and mineralized deposits on teeth (index 0 (no plaque) to 3).
Time Frame: Baseline, 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsating Toothbrush | Sonic Toothbrush | Manual Toothbrush
Number analyzed (Participants) | 28 | 30 | 24
units on a scale
  Baseline | 1.07 (0.24) | 1.19 (0.25) | 1.31 (0.27)
  1 Month | 1.11 (0.27) | 1.27 (0.40) | 1.20 (0.24)
Statistical Analysis 1: Comparison: Pulsating Toothbrush vs Sonic Toothbrush vs Manual Toothbrush; Compare groups with respect to plaque level after 30 days; Test type: Other; p = 0.1561, ANOVA — p < 0.05 considered significant

2. Primary Outcome: Gingival Index
Description: gingival index as evaluated by Silness-Loe Index, Range 0-3: Score 0 = Normal gingiva. Score 1 = Mild inflammation - slight change in color, slight edema. No bleeding on probing.
  Score 2 = Moderate inflammation - redness, edema, glazing. Bleeding on probing. Score 3 = Severe inflammation - marked redness and edema, ulceration. Tendency toward spontaneous bleeding.
Time Frame: Baseline, 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual Toothbrush | Sonic Toothbrush | Pulsating Toothbrush
Number analyzed (Participants) | 28 | 30 | 24
units on a scale
  Baseline | 0.42 (0.41) | 0.35 (0.41) | 0.36 (0.39)
  1 Month | 0.22 (0.16) | 0.16 (0.16) | 0.14 (0.13)
Statistical Analysis 1: Comparison: Manual Toothbrush vs Sonic Toothbrush vs Pulsating Toothbrush; Compare groups with respect to Gingival scores at 30 days; Test type: Other; p = 0.2161, ANOVA — p < 0.05 considered significant

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Manual Toothbrush | Sonic Toothbrush | Pulsating Toothbrush
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03416985/Prot_SAP_000.pdf